CLINICAL TRIAL: NCT06097117
Title: Molecular Methods for Identifying Bacteria in Lower Respiratory Tract Specimens Among Patients With Pneumonia by Multiplex PCR
Brief Title: Role of Multiplex PCR in CAP
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Asmaa Saleh Mousa Ali, Resident doctor at Chest department, Assiut University
Other Study IDs: role of multiplex PCR in CAP
Record Dates: First submitted 2023-09-01; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Community-acquired Pneumonia
MeSH Terms: conditions — Community-Acquired Pneumonia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- one group undergoes multiplex PCR: treatment will be started according targeted antibiotics
  Interventions: Diagnostic Test: MultiplexPCR
- the other group undergoes simple culture and sensitivity: empirical antibiotics will be started until results appear and according results ,treatment will be completed or shifted to another treatment or be narrowed ,later on detect outcome of both groups.

INTERVENTIONS:
Diagnostic Test: MultiplexPCR — PCR is a simple, yet elegant, enzymatic assay, which allows for the amplification of a specific DNA fragment from a complex pool of DNA.. Only trace amounts of DNA are needed for PCR to generate enough copies to be analyzed using conventional laboratory methods. For this reason, PCR is a sensitive assay.
  Groups: one group undergoes multiplex PCR

SUMMARY:
1. role of multiplex PCR in early identifying bacteria in patients with lower respiratory tract infection.
2. effect of early starting targeted antibiotics on outcome

DETAILED DESCRIPTION:
Pneumonia remains a worldwide health problem with a high rate of morbidity and mortality. Identification of microbial pathogens which cause pneumonia is an important area for optimum clinical management of pneumonia patients and is a big challenge for conventional microbiological methods. The development and implementation of molecular diagnostic tests for pneumonia has been a major advance in the microbiological diagnosis of respiratory pathogens in recent years. Targeted antibiotic selection and more effective de-escalation and improved stewardship for pneumonia patients.

PCR is a simple, yet elegant, enzymatic assay, which allows for the amplification of a specific DNA fragment from a complex pool of DNA.. Only trace amounts of DNA are needed for PCR to generate enough copies to be analyzed using conventional laboratory methods. For this reason, PCR is a sensitive assay.

Each PCR assay requires the presence of template DNA, primers, nucleotides, and DNA polymerase .The DNA polymerase is the key enzyme that links individual nucleotides together to form the PCR product. The nucleotides include the four bases - adenine, thymine, cytosine, and guanine (A, T, C, G) - that are found in DNA. These act as the building blocks that are used by the DNA polymerase to create the resultant PCR product. The primers in the reaction specify the exact DNA product to be amplified. The primers are short DNA fragments with a defined sequence complementary to the target DNA that is to be detected and amplified. These serve as an extension point for the DNA polymerase to build on.There are multiple advantages to PCR. First, it is a simple technique to understand and to use, a nd it produces results rapidly. It is a highly sensitive technique with the potential to produce millions to billions of copies of a specific product for sequencing, cloning, and analysis. Although PCR is a valuable technique, it does have limitations. Because PCR is a highly sensitive technique, any form of contamination of the sample by even trace amounts of DNA can produce misleading results . In addition, in order to design primers for PCR, some prior sequence data is needed. Therefore, PCR can only be used to identify the presence or absence of a known pathogen or gene

ELIGIBILITY:
Inclusion Criteria:

* male and female
* Age >18 years Old

Adult patients were included if they fulfilled:

* radiographic and clinical criteria.
* Radiographic findings included chest imaging with an airspace opacity, lobar consolida-tion, or interstitial opacities
* new or worsening compared to available baseline. In addition, at least 2 of the following clinical criteria had to be fulfilled:

  1. reported or documented fever > 37.5
  2. new worsening productive cough or increase in respiratory secretions in intubated patients
  3. pleuritic chest pain 4) new/worsening dyspnea or hypoxia, defined as documented blood oxygen saturation <92%.

     Exclusion Criteria:

     Patients under 18 years old. Patients who refuse to participate in the study

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with CAP will divided in two groups (1:1), one group undergoes multiplex PCR and treatment will be started according targeted antibiotics, the other group undergoes simple culture and sensitivity and empirical antibiotics will be started until results appear and according results ,treatment will be completed or shifted to another treatment or be narrowed ,later on detect outcome of both groups.
  Sample Size Calculation: 66 cases
Sampling Method: Non-Probability Sample
Enrollment: 66 (Estimated)
Dates: Start 2023-11-01 (Estimated); Primary Completion 2024-10-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
detect Antimicrobial therapy duration in CAP in comparison in both groups | 1 year
  Antimicrobial therapy duration in patients with CAP in comparison of two groups
detect clinical improvement in both groups | 1 year
  detection of clinical improvement in both groups (subsided of bronchial symptoms as productive cough ,colored sputum, relieve of dysnea and pleuritic chest pain , subsided of fever

REFERENCES:
- See also: . Timsit J-F, Bassetti M, Cremer O, et al. Rationalizing antimicrobial therapy in the ICU: a narrative review. Intensive Care Med. 2019;45(2):172-89 — https://doi.org/10.1007/s00134-019-05520-5
- See also: . Peiffer-Smadja N, Rawson TM, Ahmad R, et al. Machine learning for clinical decision support in infectious diseases: a narrative review of current applications. Clin Microbiol Infect Published online September 17. 2019 — https://doi.org/10.1016/j.cmi.2019.09.009